CLINICAL TRIAL: NCT06396741
Title: Determination of Biomechanical Changes in the Quadriceps Muscle After Dry Needling Treatment
Brief Title: Changes in the Quadriceps Muscle After Dry Needling Treatment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Daniel Pecos Martín (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Daniel Pecos Martín, Professor, University of Alcala
Organization: University of Alcala (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CEID/2022/5/092
Record Dates: First submitted 2024-04-25; First posted 2024-05-02 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Muscle Tightness; Muscle Strain
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Quadriceps muscle dry needling (Experimental): The Quadriceps muscle will be punctured with ultrasound control
  Interventions: Other: The quadriceps muscle will be punctured with ultrasound control

INTERVENTIONS:
Other: The quadriceps muscle will be punctured with ultrasound control — With the subject in the supine position, the quadriceps muscle will be shown by ultrasound. Subsequently, a dry needling technique will be performed at the most hyperalgesic point using ultrasound control.

SUMMARY:
The present study aims to examine the mechanical changes following dry needling of the quadriceps muscle.

To this end, structural and mechanical changes in quadriceps muscle activity will be measured using M-mode ultrasound.

The quadriceps muscle strength will also be assessed with dynamometry. In addition, the knee joint range will be checked by means of a goniometry procedure.

The subjects will be assessed before and after the application of a dry needling technique on the quadriceps muscle to determine possible changes in the measured variables.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject.

Exclusion Criteria:

* Low back pain
* Hip pain
* Sciatica
* Belenophobia
* Be medicated with anticoagulants
* Knee surgery
* Knee osteoarthritis
* Fibromyalgia
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Muscle thickness | before and after one week. The muscle thinckness will be measurement in centimeters
  Muscle thickness and echo intensity, an indicator of muscle quality, are related to muscle strength, physical function, and muscle mass measured using echographs ultrasound.It will be measured how muscle thickness changes after applying a dry needling technique

SECONDARY OUTCOMES:
Quadriceps muscle strength | before and after one week.
  The quadriceps muscle strength evaluation will be the measurement of isometric knee extension strength with a hand-held dynamometer (microFET2, Hoggan Scientific, LLC; West Jordan, UT). The maximum voluntary contraction of the quadriceps muscle will be measured. The participants completed three maximal isometric contractions, holding for approximately 3 seconds, with one minute of rest between each contraction.The value of the force will be obtained by calculating the average of the three measurements. The muscle strength wil be measurement in kilograms
knee range of motion (flexion) | before and after one week
  To measure knee flexion, bend the knee as far as you can, by sliding your foot up towards your buttocks, keeping the arms and axis of the goniometer in place, then measure. Passive Knee Flexion ROM: up to 150º, depending on the size of the leg - the limit is the calf pushing onto the back of the thigh. The knee range of motion will be measurement in degrees

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Fernandez-Carnero, PhD, Study Chair — Centro de Investigación Fisioterapia y Dolor
Locations (1):
- Centro Investigación Fisioterapia y Dolor, Alcalá de Henares, Madrid, Spain